CLINICAL TRIAL: NCT00355914
Title: A Randomized, Prospective, Double-Blind Controlled Evaluation of the Effectiveness of Lumbar Facet Joint Nerve Blocks
Brief Title: Effectiveness of Lumbar Facet Joint Nerve Blocks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pain Management Center of Paducah (Other)
Responsible Party: Principal Investigator, Laxmaiah Manchikanti, MD, CEO, Pain Management Center of Paducah
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: protocol3
Record Dates: First submitted 2006-07-24; First posted 2006-07-25 (Estimated); Results first posted 2013-11-26 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-09

CONDITIONS: Low Back Pain
Keywords: Lumbar Facet Joint Nerve Block
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 Without Steroids (Active Comparator): Lumbar Facet Joint Nerve Block with Local Anesthetic (0.5 mL of 0.25% Bupivacaine with/without 0.5 mL of Sarapin)
  Interventions: Procedure: Lumbar Facet Joint Nerve Block
- Group 2 With Steroids (Experimental): Lumbar Facet Joint Nerve Block with Local Anesthetic (0.5 mL of 0.25% Bupivacaine with/without 0.5 mL of Sarapin) and 0.15 mg of non-particulate betamethasone)
  Interventions: Procedure: Lumbar Facet Joint Nerve Block

INTERVENTIONS:
Procedure: Lumbar Facet Joint Nerve Block — Lumbar Facet Joint Nerve Block

SUMMARY:
1. To demonstrate whether:

   i. Facet joint nerve blocks have therapeutic value beyond the duration of local anesthetic effect.

   ii. Adjuvant medications (Sarapin and Depo-steroids) provide additional relief of lumbar facet joint pain when used with facet joint nerve blocks.
2. To demonstrate whether or not there are clinically significant improvements in function of patients who receive lumbar facet joint nerve block with or without Sarapin and Depo-steroids (Group II) compared to patients randomized to Group I who receive only local anesthetic blocks.
3. To determine the adverse event profile in both groups.

DETAILED DESCRIPTION:
Primary Outcome Measure(s) To demonstrate a clinically significant difference between the patients treated with adjuvants and those patients randomized to Group I in the pain status, physical, and psychological status and pain at 3, 6, 12, 18and 24 months post treatment.

ELIGIBILITY:
Inclusion Criteria:

* Positive for facet joint pain with comparative local anesthetic blocks

Candidates are over 18 years of age

Subjects with a history of chronic, function limiting low back pain of at least six months in duration Subjects who are able to give voluntary, written informed consent to participate in this investigation Subjects who, in the opinion of the Investigator, are able to understand this investigation, co-operate with the investigational procedures and are willing to return to the center for all the required post-operative follow-ups The subject has not had recent surgical procedures within the last three months.

Exclusion Criteria:

* Negative or false-positive response to controlled comparative local anesthetic blocks

Narcotic use of greater than Hydrocodone 100 mg/day, Methadone 80 mg or Morphine 100 mg, or dose equivalent

Uncontrolled major Depression or uncontrolled psychiatric disorders

Uncontrolled or acute medical illnesses including coagulopathy, renal insufficiency, chronic liver dysfunction, progressive neurological deficit, urinary sphincter dysfunction, infection, increased intercranial pressure, pseudotumor cerebri, intercranial tumors, unstable angina, and severe chronic obstructive pulmonary disease.

Chronic severe conditions that could interfere with the interpretations of the outcome assessments for pain and bodily function

Women who are pregnant or lactating

Subjects who have participated in a clinical study with an investigational product within 30 days of enrollment

Patients with multiple complaints involving concomitant hip osteoarthritis, will not be amenable to study due to the overlap of pain complaints.

Inability to achieve appropriate positioning and inability to understand informed consent and protocol History of adverse reaction to local anesthetic or anti-inflammatory drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2003-08; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laxmaiah Manchikanti, MD, Principal Investigator — Ambulatory Surgery Center
Locations (1):
- Ambulatory Surgery Center, Paducah, Kentucky, United States

REFERENCES:
- [Result] Manchikanti L, Singh V, Falco FJ, Cash KA, Pampati V. Evaluation of lumbar facet joint nerve blocks in managing chronic low back pain: a randomized, double-blind, controlled trial with a 2-year follow-up. Int J Med Sci. 2010 May 28;7(3):124-35. doi: 10.7150/ijms.7.124. PMID 20567613
- [Result] Manchikanti L, Singh V, Falco FJ, Cash KA, Pampati V. Lumbar facet joint nerve blocks in managing chronic facet joint pain: one-year follow-up of a randomized, double-blind controlled trial: Clinical Trial NCT00355914. Pain Physician. 2008 Mar-Apr;11(2):121-32. PMID 18354721
- [Result] Manchikanti L, Manchikanti KN, Manchukonda R, Cash KA, Damron KS, Pampati V, McManus CD. Evaluation of lumbar facet joint nerve blocks in the management of chronic low back pain: preliminary report of a randomized, double-blind controlled trial: clinical trial NCT00355914. Pain Physician. 2007 May;10(3):425-40. PMID 17525777
- See also: Evaluation of lumbar facet joint nerve blocks in managing chronic low back pain: a randomized, double-blind, controlled trial with a 2-year follow-up. — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC2880841/pdf/ijmsv07p0124.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period lasted from November 2003 to July 2006.
Groups:
- Group 1 Without Steroids: Lumbar Facet Joint block with Local Anesthetic (0.5 mL of 0.25% Bupivacaine with/without 0.5 mL of Sarapin)
- Group II With Steroids: Lumbar Facet Joint block with Local Anesthetic (0.5 mL of 0.25% Bupivacaine with/without 0.5 mL of Sarapin) and Steroids (0.15 mg of non-particulate betamethasone)
Period: Overall Study
Arm/Group | Group 1 Without Steroids | Group II With Steroids
Started | 60 | 60
Completed | 60 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1 Without Steroids: Lumbar Facet Joint Nerve Blocks Local anesthetic without steroids
- Group II With Steroids: Lumbar Facet Joint Nerve Blocks Local anesthetic with steroids
- Total: Total of all reporting groups
Arm/Group | Group 1 Without Steroids | Group II With Steroids | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 51 | 53 | 104
  >=65 years | 9 | 7 | 16
Age Continuous [Mean (Standard Deviation); unit: years] | 47 (15) | 46 (17) | 46.7 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 33 | 72
  Male | 21 | 27 | 48
Region of Enrollment [Number; unit: participants]
  United States | 60 | 60 | 120

OUTCOME MEASURES:

1. Primary Outcome: Average Numeric Rating Scale
Description: Numeric rating scale represented 0 with no pain and 10 with the worst pain imaginable.
Time Frame: Baseline, 3, 6, 12, 18, and 24 months post-treatment
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Group I: Local anesthetic without steroids
- Group II: Local anesthetic with steroids
Arm/Group | Group I | Group II
Number analyzed (Participants) | 60 | 60
units on a scale
  Baseline | 8.2 (0.8) | 7.9 (1.0)
  3 months | 3.8 (1.3) | 3.5 (1.1)
  6 months | 3.6 (1.5) | 3.3 (0.8)
  12 months | 3.7 (1.7) | 3.5 (1.1)
  18 months | 3.5 (1.5) | 3.3 (1.0)
  24 months | 3.5 (1.5) | 3.2 (0.9)
Statistical Analysis 1: Comparison: Group I vs Group II; compared baseline, 3, 6, 12, 18, and 24 months between groups; Test type: Superiority or Other; p > 0.05, t-test, 2 sided — Results were considered statistically significant if the P value was less than 0.05

2. Primary Outcome: Oswestry Disability Index
Description: Oswestry Disability Index 2.0 (ODI): ODI score is ranged from 0 to 50. Total score is converted in to percent disability. ODI Scoring: 0% to 20% (minimal disability), 21%-40% (moderate disability), 41%-60% (severe disability), 61%-80% (crippled) and 81%-100% (may be bed bound or exaggerating their symptoms).
Time Frame: Baseline, 3, 6, 12, 18, and 24 months post-treatment.
Population: An intent-to-treat-analysis was performed on all patients utilizing the last follow-up data. Initial data were utilized in the patients who dropped out of the study without further follow-up after the first treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Group II With Steroids: Facet Joint Nerve Blocks Local anesthetic with steroids
Arm/Group | Group 1 Without Steroids | Group II With Steroids
Number analyzed (Participants) | 60 | 60
units on a scale
  Baseline | 26.6 (4.6) | 25.9 (5.0)
  3 months | 12.7 (4.7) | 13.5 (5.6)
  6 months | 12.7 (4.7) | 12.2 (5.0)
  12 months | 12.3 (4.8) | 12.0 (5.4)
  18 months | 12.1 (5.0) | 11.2 (4.9)
  24 months | 12.0 (4.9) | 11.0 (4.8)
Statistical Analysis 1: Comparison: Group 1 Without Steroids vs Group II With Steroids; baseline, 3, 6, 12, 18, and 24 months between groups; Test type: Superiority or Other; p > 0.05, t-test, 2 sided — Results were considered statistically significant if the P value was less than 0.05

ADVERSE EVENTS:
Arm/Group | Group 1 Without Steroids | Group II With Steroids
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes